CLINICAL TRIAL: NCT03934567
Title: An Open-label, Single-arm, Multi-center Phase 2 Study to Evaluate the Efficacy and Safety of Oral Histone Deacetylase (HDAC)-Inhibitor Abexinostat, as Monotherapy in Patients With Relapsed or Refractory Follicular Lymphoma (FL)
Brief Title: A Multi-Center Phase 2 Study to Evaluate Efficacy and Safety of Oral Abexinostat as Monotherapy in Patients With Relapsed or Refractory Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYN-605
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma, Follicular
Keywords: refractory; relapsed; lymph nodes
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — abexinostat

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abexinostat 80 mg bis in die (BID) (Experimental): Experimental: Abexinostat 80 mg BID
  Interventions: Drug: Abexinostat

INTERVENTIONS:
Drug: Abexinostat — Abexinostat tablets

SUMMARY:
An open-label, single-arm, multi-center phase 2 study to evaluate the efficacy and safety of oral histone deacetylase (HDAC)-inhibitor abexinostat, as monotherapy in patients with relapsed or refractory follicular lymphoma (FL)

DETAILED DESCRIPTION:
This is an open-label, single-arm, two-stage, multi-center, phase 2 study in patients with relapsed/refractory follicular lymphoma (FL) who have received at least two prior standard therapy lines.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy ≥ 3 months
2. Histologically confirmed grade 1, 2, or 3a follicular lymphoma (FL)
3. Have received at least two prior standard therapy lines including anti- cluster of differentiation antigen (anti-CD20) antibody and cytotoxic therapy for follicular lymphoma (FL)
4. Confirmed to be unresponsive to the last line of therapy (have stable disease or disease progression during treatment),or have disease progression following the last line of therapy
5. Have at least one radiologically measurable lymph node or extranodal lymphoid malignant lesion as assessed by computed tomography (CT) or magnetic resonance imaging (MRI);
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
7. Meet various hematological, liver function and renal function lab parameters

Exclusion Criteria:

1. Histologically confirmed grade 3b follicular lymphoma, or transformed diffuse large B-cell lymphoma (DLBCL)
2. Current or history of central nervous system (CNS) lymphoma;
3. Toxicity not yet recovered from previous anti-tumor therapies
4. Uncontrolled systemic infections or infections requiring intravenous antibiotics
5. Have previously treated by abexinostat or other histone deacetylase (HDAC) inhibitors;
6. Have received steroid hormone within 7 days, chemotherapy, targeted therapy within 28 days, radiotherapy within 14 days, anti-cancer antibody therapies within 28 days
7. Unable to swallow tablets, or presence of significant functional gastrointestinal disorders that may affect the oral administration and absorption of the study drug
8. Have received autologous stem cell transplant within 3 months before the first dose, or allogeneic stem cell transplant within 6 months before the first dose
9. Presence of active graft-versus-host disease
10. Have undergone a major surgery within 28 days
11. Evidence of possible human immunodeficiency virus (HIV) infection or hepatitis C virus (HCV) infection
12. Have cardiac impairment as defined per protocol
13. Have prior history of malignancies other than follicular lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical effect of abexinostat on objective response rate as assessed by an independent central imaging review | up to 56 days
  Objective response rate (ORR), defined as the proportion of patients who have completed response (CR) or partial response (PR) as assessed by an Independent Central Imaging Review

SECONDARY OUTCOMES:
Objective Response | up to 56 days
  Objective response rate (ORR) as assessed by the investigator
Progression-free survival | Up to 2 years
  Progression-free survival (PFS), defined as the time from the initiation of treatment to disease progression or death as assessed by the Independent Central Imaging Review and the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai SHI, Prof, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (26):
- China (26):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Medical University Union Hospital, Fuzhou
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - Sun Yai-Sen Memorial Hospital, Sun Yai-Sen University, Guangzhou
  - Nanfang Hospital, Guangzhou
  - Hainan General Hospital, Hainan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medical, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - The First Hospital of Lanzhou University, Lanzhou
  - Linyi Cancer Hospital, Linyi
  - Nantong Tumor Hospital, Nantong
  - Shanghai Sixth people's hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - The Forth Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin People's Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No